CLINICAL TRIAL: NCT01869660
Title: Shared Decision Making for Patients With First-admission Schizophrenia: a Randomized Controlled Trial
Brief Title: Shared Decision Making for Patients With First-admission Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yokohama City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDMS-S
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: First hospitalization
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shared Decision Making (Experimental): The present SDM intervention is based on principles derived from previous randomized controlled trials of SDMs. SDM meetings comprise at least 4 weekly 20 minutes sessions. Meetings have at least three professionals: a case manager (psychiatrists or nurses), a primary doctor, and a nurse/social worker. The focus of the meeting is to empower patients to discuss their attitudes and preferences toward treatments.
  Interventions: Behavioral: Shared Decision Making
- Usual Care (No Intervention): Patients with no special program about decision making.

INTERVENTIONS:
Behavioral: Shared Decision Making — The focus of the SDM is to empower patients to discuss their attitudes and preferences toward treatments.
  Arms: Shared Decision Making

SUMMARY:
To determine whether shared decision making (SDM) intervention improves patient satisfaction in patients with first-admission schizophrenia compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an acute care psychiatric ward.
* Diagnosed with schizophrenia (ICD-10 codes: F20-F29)
* Aged 16 to 65 years old at admission
* No prior experience of psychiatric admission (first-admission)

Exclusion Criteria:

* Diagnosed with moderate to severe mental retardation
* Diagnosed with organic mental disorders (ICD10 codes: F00-F09)
* Having poor Japanese language skill
* Severe conceptual disorganization as measured by brief psychiatric rating scale of 5 or more.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction as measured by the Japanese version of the Client Satisfaction Questionnaire (CSQ-8) | Within 7days before the date of discharge

SECONDARY OUTCOMES:
Attitude toward medication as measured by the Japanese version of the Drug Attitude Inventory (DAI-10) | Within 7days before the date of discharge
Treatment continuation as measured by the rate of outpatient attendance during the 30 days | 6 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Hirayasu, PhD, Study Chair — Department of Psychiatry, Yokohama City University School of Medical
Locations (1):
- Numazu Chuou Hospital, Numazu, Shizuoka, Japan

REFERENCES:
- [Derived] Ishii M, Okumura Y, Sugiyama N, Hasegawa H, Noda T, Hirayasu Y, Ito H. Feasibility and efficacy of shared decision making for first-admission schizophrenia: a randomized clinical trial. BMC Psychiatry. 2017 Feb 6;17(1):52. doi: 10.1186/s12888-017-1218-1. PMID 28166757
- [Derived] Ishii M, Okumura Y, Sugiyama N, Hasegawa H, Noda T, Hirayasu Y, Ito H. Efficacy of shared decision making on treatment satisfaction for patients with first-admission schizophrenia: study protocol for a randomised controlled trial. BMC Psychiatry. 2014 Apr 14;14:111. doi: 10.1186/1471-244X-14-111. PMID 24725910